CLINICAL TRIAL: NCT04796532
Title: Home Based or Traditional Class HIIT in Overweight Women: Effects on Physical Activity, Body Composition and Cardio Respiratory Fitness. A 3-arm Randomized Control Trial.
Brief Title: Home Based or Traditional Class HIIT in Overweight Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Évora (Other)
Collaborators: Raimundo, Armando, PhD (Unknown); Bravo, Jorge, PhD (Unknown); Mota, Jorge, PhD, University of Porto (Unknown)
Responsible Party: Principal Investigator, João Luis Fernandes do Carmo, Doctoral Student, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21016
Record Dates: First submitted 2021-02-24; First posted 2021-03-15 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Overweight or Obesity
Keywords: High Intensity Training; Exercise; Home-based; Overweight; Women
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: 3 arm parallel groups
Who Masked: Participant
Masking Description: The participants will be randomized and alllocated in one of the three groups (control or experimental HIIT Homebased or experimental HIIT traditional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention. The control group will maintain their normal physical and dietary activity.
- Homebased HIIT (Experimental): 16-week exercise program with HIIT with a frequency of 3 days/week. The Homebased HIIT group participants will attend HIIT workout sessions supervised by a specialised instructor via a videoconference application. This group will have 16 week follow-up.
  Interventions: Other: Home based HIIT
- Traditional HIIT (Experimental): 16-week exercise program with HIIT with a frequency of 3 days/week. The Traditional-HIIT group participants will attend presential HIIT workout sessions supervised. This group will have 16 week follow-up.
  Interventions: Other: Traditional HIIT

INTERVENTIONS:
Other: Home based HIIT — Intervention will consist in a 16-week exercise program with HIIT with a frequency of 3 days/week. The Home-HIIT group participants will attend HIIT workout sessions supervised by a specialised instructor via a videoconference application. Every HIIT workout session will have a 10 minutes' warm-up, followed by an 8/12/16/20 minutes of HIIT (stages of physical adaptation every 4 weeks) training and 5 minutes' cool-down. Tabata method will be used with eight sets of 20 seconds of exercise bouts separated by 10 seconds rest, in 2 to 5 blocks. The intervention will have four stages of physical adaptation.
  This group will have a follow-up period of 16 weeks.
  Arms: Homebased HIIT
Other: Traditional HIIT — Intervention will consist in a 16-week exercise program with HIIT with a frequency of 3 days/week. The Traditional HIIT group participants will attend a group HIIT workout sessions supervised by a specialised instructor in a sport facility. Every HIIT workout session will have a 10 minutes' warm-up, followed by an 8/12/16/20 minutes of HIIT (stages of physical adaptation every 4 weeks) training and 5 minutes' cool-down. Tabata method will be used with eight sets of 20 seconds of exercise bouts separated by 10 seconds rest, in 2 to 5 blocks. The intervention will have four stages of physical adaptation.
  This group will have a follow-up period of 16 weeks.
  Arms: Traditional HIIT

SUMMARY:
The present protocol aims to evaluate the effect of two different 16-week High-intensity interval training (HIIT) programs on daily physical activity, body composition, cardiorespiratory fitness, eating behaviour, enjoyment and quality of life in overweight women. Methods: Ninety overweight women (25 - 50 years old) with a body mass index ≥ 25 kg/m2 will be randomly assigned to three groups of 30 participants: a remote home-based HIIT intervention group; a traditional HIIT intervention group; and a non-exercise control group. Both intervention groups will undergo a 16-week progressive HIIT program following the Tabata method. Participants will be assessed at baseline, 4th, 8th, and after 16-week for physical activity, body composition, cardiorespiratory fitness, eating behaviour, enjoyment and quality of life. The study will have a 16-week follow-up post intervention. Results: The participant's enrolment will begin in December 2021, and investigators will anticipate the study completion by the mid of 2022. Conclusions: The HIIT programs might have beneficial effects on daily physical activity, body composition, cardiorespiratory fitness and overall quality of life in overweight women. Moreover, it might be a more enjoyable form of exercise, once it is performed faster than other exercise forms. As a beneficial side effect, these healthy behaviours might have a favourable impact on women's eating behaviours. This study results are expected to add health and well-being professionals' evidence-based knowledge to create strategies and design home-based exercise interventions.

DETAILED DESCRIPTION:
Methods Trial design: The study will be a 3-arm Randomized Controlled Trial, in which a similar number of participants will be assigned to three groups: a supervised remote home-based HIIT intervention group (Home-HITT), or a presential a supervised traditional HIIT intervention group (Traditional-HIIT), and a non-exercise control group (CG). The study will have a 32-week duration and will be carried out in Portugal. This RCT will be "single-blind".

This study has been designed according to CONSORT statement for clinical trials. This RCT will apply the "intention-to-treat principle".

Dose rationale: The CG participants will maintain their usual physical and dietary activity. Nevertheless, after the 16-week intervention, participants selected to the CG will have the chance to receive the same 16-week HIIT program. Both interventions will consist of a 16-week exercise program with HIIT with a frequency of 3 days/week. The Home-HIIT group participants will attend HIIT workout sessions supervised by a specialised instructor via a videoconference application, while the Traditional-HIIT group participants will attend HIIT workout sessions supervised in person by the same instructor. Every HIIT workout session will have a 10 minutes' warm-up, followed by an 8/12/16/20 minutes of HIIT training and 5 minutes' cool-down. The intervention will have a type of HIIT program called the Tabata method once it can be performed in home-based programs. Tabata training method has been defined as a HIIT with submaximal effort performed at 80-95% of maximal heart rate.

Tabata method uses eight sets of 20 seconds of exercise bouts separated by 10 seconds rest, in 2 to 5 blocks. It seems that this method is demanding for ordinary adults so it will have four stages of physical adaptation.

Before each session, all participants in the intervention groups will receive a class reminder through a short message service (SMS). After each session, all participants will also receive an SMS with positive reinforcement about their exercise session participation. In order to compensate for possible absences, extra classes will be given. The 16 weeks intervention period was chosen because evidence shows that this period is sufficient to evidence changes in PA levels. Guidelines suggest the need to accumulate 75 min/week of vigorous-intensity PA. Despite the guidelines, this exercise protocol will be characterized by progression in both exercise intensity and volume because the investigators will be handling sedentary and overweight women.

The present study will have a follow-up period of 16 weeks. During this period, it is necessary to verify the study variables' evolution.

Selection and Withdrawal of Subjects: Participants in this study will be volunteers recruited through Health Centers Portimão, Lagoa and Lagos (Algarve, Portugal) and through promotional flyers placed in region´s local councils. All the participants will be informed of the procedures of the study before signing the informed consent form.

Subject Withdrawal: Individuals will be removed from the study when the following situations are verified: i) medical indication; ii) prolonged illness during the study or injury incapacitating to continue the study; iii) show willingness to leave the study. Participants may be replaced if the withdrawal happens before the intervention starts.

Discontinuation: The study should be interrupted if it is found that the application of the HIIT exercise program is at the origin of the participants physical and/or psychological problems. There will also be an interruption of the study if it is found that the participant initiated a physical exercise program parallel to the study.

Sample size Determination: To determine a priori the sample size, investigators used G*Power (version 3.1.9.7). The sample size was determined by the study's primary objective (effect of the intervention on PA, body composition and cardiovascular health). Based on a large effect size of 0.80 (Cohen's f), performing a sample size calculation for repeated measures analysis of variance with an expectable correlation of 0.50 between measurements, alfa of 0.05 and 85% of power, a total sample size of 60 women will be needed.

Once the investigators have two experimental groups, the aim is to have 90 women in this study.

Statistical Analysis SPSS (StatisticalPackage for the SocialSciences) software, version 27.0, IBM Windows will be used.

Regarding the procedures for sample distribution characterization's, the mean, standard deviation and amplitude of the distribution (min. value and max. value) will be determined. To determine data normality, the investigators will use the Kolmogorov-Smirnov analysis. Parametric statistics will be applied if data is normally distributed. One-way ANOVA will be used for comparisons of the three groups on all outcome's variables. To determine the relation between the independent measures, the investigators will use a two-way ANOVA. If there are significant differences between the different groups, the Bonferroni Post-hoc test will determine significance levels. In this study, the investigators will use a p-value of 0.05.

Randomization: In order to minimize selection bias, stratified randomization will be carried out when allocating individuals to the experimental and control groups, thus maintaining identical characteristics in both groups This stratification will be carried out based on age, sex and ethnicity.

Instruments: For the present study, participants will be evaluated before the intervention in the 4th ,8th and 16th week of the intervention. After that, participants will be evaluated in the 32nd week for follow-up to analyse the possible effect of detraining. Assessments will be performed through the following instruments:

1. Sociodemographic questionnaire - Questionnaire made for the study with questions about age, sex;
2. Anthropometry and Body Composition - Stature and weight will be evaluated to calculate body mass index. Weight and statures will be measured to the nearest 0.1Kg and 0.1cm correspondingly (calibrated weighing-machine and stadiometer). For the body mass index calculation, weight in kilo-grams will be divided by the height in squared meters. The criteria for defining excess weight and obesity proposed by World Health Organization. The waist circumference will be recorded using a non-elastic measuring tape, which is placed horizontally above the top of the iliac crest. This measurement should be performed with a tense tape without compressing the skin and at the end of exhalation. It will be assessed % fat mass, bone mass and muscle mass with a bioimpedance weighing-machine electric model Tanita BC601. Before the test, the participants will be told to lie down in a supination position to ensure good blood circulation;
3. Blood Pressure (BP) - The BP will be assessed using electronic BP device OMRON M2 (13) according to validation protocols;
4. PA Questionnaire - For measuring PA, by questionnaire it will be used International Physical Activity Questionnaire - Long Version (IPAQ);
5. Daily PA - Objectively measured daily PA will be assessed through accelerometers, using the Model ActiGraph GT3X+ (Pensacola, USA), triaxial accelerometer, supported by the ActiLife Software. ActiGraf models have been widely used in research, and it is estimated that more than 50% of the research using accelerometry uses this brand. Participants will use the accelerometer for seven consecutive days, during the day and night (night sleep), except for activity involving water (e.g., swimming) or contact (e.g., combat sports). The devices will be placed in the hip because it seems to be more effective in classifying the intensity of PA and the movement patterns. The accelerometer will be programmed for 60 seconds epoch length. Each day will only be considered when recording at least 600 minutes of activity, i.e., 10 hours. The daily time spent in light, moderate and vigorous-intensity activities will be calculated;
6. Exercise intensity - Investigators will monitor exercise intensity with the perceived exertion Borg Scale. This scale has been used in RCT with HIIT;
7. Cardiorespiratory Fitness (CRF) - To assess VO2max the Chester Step Test will be used. This field test proved to be reliability to estimate CRF and has been used in controlled trials with the overweight population;
8. Enjoyment - To measure the enjoyment, the investigators will use Portuguese version of the the Physical Activity Enjoyment Scale (PACES);
9. Quality of life - To assess the quality of life it will be used the Portuguese version of the SF-36 Questionnaire. This questionnaire evaluates 8 dimensions: physical function, physical performance, physical pain, general health, mental health, emotional performance, social function and vitality;
10. Eating Behaviour - The eating behaviour will be assessed through the Portuguese version of the Three-Factor Eating Questionnaire - R21 (TFEQ - R21) questionnaire, consisting of 21 items and three subscales: cognitive restraint, uncontrolled eating and emotional eating;
11. Satisfaction with the study - A satisfaction Likert-scale questionnaire that the participants should fill out, aims to assess the satisfaction with the exercise classes. The Likert-scale questionnaire will be created for this purpose.

Timing: According to the inclusion/exclusion criteria mentioned, the participants will be assessed to be eligible to participate in the study. In December 2021, participants will be randomized and allocated in three different groups (CG, Home HIIT and Class HIIT). The intervention will begin in December 2021 and end in September 2022. The close-out of the study will be in September.

ELIGIBILITY:
Inclusion Criteria:

* female individuals aged between 25 and 50 years old, at the time of selection;
* have a BMI equal to or greater than 25kg/m2;
* have the ZOOM application (San Jose, USA) and a 2x2m2 space at home for the practice of HIIT;
* who present, in their own form, authorized consent to participate in the referred study. Only one person per household will be allowed to be included.

Exclusion Criteria:

* having any health problem and/or condition that limit the implementation of an HIIT program;
* taking medication that influences the variables to be studied;
* being involved in any type of exercise intervention/program;
* being in pre-menopause or menopause period.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Overweight women between 25 and 50 years old.
Enrollment: 90 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline, between and within groups comparison, in Physical activity. | 0,4,8,16,32 weeks
  Objectively measured daily physical activity will be assessed through accelerometers.
Change from Baseline, between and within groups comparison, in Cardiorespiratory fitness. | 0,4,8,16,32 weeks
  To assess VO2max the Chester Step Test will be used.
Change from Baseline, between and within groups comparison, in percentage of fat mass. | 0,4,8,16,32 weeks
  It will be assessed % fat mass with a bioimpedance weighing machine electric model Tanita BC601.
Change from Baseline, between and within groups comparison, in bone mass. | 0,4,8,16,32 weeks
  It will be assessed bone mass with a bioimpedance weighing machine electric model Tanita BC601. The bone mass will be reported in kilograms.
Change from Baseline, between and within groups comparison, in muscle mass. | 0,4,8,16,32 weeks
  It will be assessed muscle mass with a bioimpedance weighing machine electric model Tanita BC601. The muscle mass will be reported in kilograms.
Change from Baseline, between and within groups comparison, in body mass index (BMI). | 0,4,8,16,32 weeks
  Weight and height will be measured to the nearest 0.1kg and 0.1cm correspondingly. For BMI, weight in kilograms will be divided by height in squared meters (kg/m2).

SECONDARY OUTCOMES:
Change from Baseline, between and within groups comparison, in Quality of Life | 0,4,8,16,32 weeks
  To assess the quality of life it will be used the Portuguese version of the SF-36 Questionnaire
Change from Baseline, between and within groups comparison, in Eating Behaviour | 0,4,8,16,32 weeks
  The eating behaviour will be assessed through the Portuguese version of the Three-Factor Eating Questionnaire - R21
Change from Baseline, between and within groups comparison, in Enjoyment | 0,4,8,16,32 weeks
  To measure the enjoyment it will use Portuguese version of the the PACES scale. This is a 8-item scale. Each item has a 7-point Likert scale (1= unpleasurable; 7= pleasurable).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Mota, PhD, Study Director — Universidade do Porto; Armando Raimundo, PhD, Study Director — Universidade de Evora

IPD SHARING:
Plan to Share IPD: Yes
Yes. We will publish the protocol and study results.
Supporting Information: ICF
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Asmar R, Khabouth J, Topouchian J, El Feghali R, Mattar J. Validation of three automatic devices for self-measurement of blood pressure according to the International Protocol: The Omron M3 Intellisense (HEM-7051-E), the Omron M2 Compact (HEM 7102-E), and the Omron R3-I Plus (HEM 6022-E). Blood Press Monit. 2010 Feb;15(1):49-54. doi: 10.1097/MBP.0b013e3283354b11. PMID 20032779
- [Background] Baptista F, Santos DA, Silva AM, Mota J, Santos R, Vale S, Ferreira JP, Raimundo AM, Moreira H, Sardinha LB. Prevalence of the Portuguese population attaining sufficient physical activity. Med Sci Sports Exerc. 2012 Mar;44(3):466-73. doi: 10.1249/MSS.0b013e318230e441. PMID 21844823
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Dekkers JC, van Wier MF, Ariens GA, Hendriksen IJ, Pronk NP, Smid T, van Mechelen W. Comparative effectiveness of lifestyle interventions on cardiovascular risk factors among a Dutch overweight working population: a randomized controlled trial. BMC Public Health. 2011 Jan 24;11(1):49. doi: 10.1186/1471-2458-11-49. PMID 21261935
- [Background] Doak CM, Wijnhoven TM, Schokker DF, Visscher TL, Seidell JC. Age standardization in mapping adult overweight and obesity trends in the WHO European Region. Obes Rev. 2012 Feb;13(2):174-91. doi: 10.1111/j.1467-789X.2011.00943.x. Epub 2011 Nov 7. PMID 22060052
- [Background] Duarte PAS, Palmeira L, Pinto-Gouveia J. The Three-Factor Eating Questionnaire-R21: a confirmatory factor analysis in a Portuguese sample. Eat Weight Disord. 2020 Feb;25(1):247-256. doi: 10.1007/s40519-018-0561-7. Epub 2018 Aug 28. PMID 30168033
- [Background] Ellis K, Kerr J, Godbole S, Lanckriet G, Wing D, Marshall S. A random forest classifier for the prediction of energy expenditure and type of physical activity from wrist and hip accelerometers. Physiol Meas. 2014 Nov;35(11):2191-203. doi: 10.1088/0967-3334/35/11/2191. Epub 2014 Oct 23. PMID 25340969
- [Background] Fabre N, Lhuisset L, Bernal C, Bois J. Effect of epoch length on intensity classification and on accuracy of measurement under controlled conditions on treadmill: Towards a better understanding of accelerometer measurement. PLoS One. 2020 Jan 24;15(1):e0227740. doi: 10.1371/journal.pone.0227740. eCollection 2020. PMID 31978093
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part II --Validation tests]. Acta Med Port. 2000 May-Jun;13(3):119-27. Portuguese. PMID 11026151
- [Background] Forberger S, Reisch L, Kampfmann T, Zeeb H. Nudging to move: a scoping review of the use of choice architecture interventions to promote physical activity in the general population. Int J Behav Nutr Phys Act. 2019 Sep 3;16(1):77. doi: 10.1186/s12966-019-0844-z. PMID 31481090
- [Background] Foster C, Farland CV, Guidotti F, Harbin M, Roberts B, Schuette J, Tuuri A, Doberstein ST, Porcari JP. The Effects of High Intensity Interval Training vs Steady State Training on Aerobic and Anaerobic Capacity. J Sports Sci Med. 2015 Nov 24;14(4):747-55. eCollection 2015 Dec. PMID 26664271
- [Background] Frimpong E, Dafkin C, Donaldson J, Millen AME, Meiring RM. The effect of home-based low-volume, high-intensity interval training on cardiorespiratory fitness, body composition and cardiometabolic health in women of normal body mass and those with overweight or obesity: protocol for a randomized controlled trial. BMC Sports Sci Med Rehabil. 2019 Dec 30;11:39. doi: 10.1186/s13102-019-0152-6. eCollection 2019. PMID 31893126
- [Background] Gillman AS, Stevens CJ, Bryan AD. Women's exercise identity increases after a 16-week exercise RCT and is linked to behavior maintenance at follow-up. Psychol Sport Exerc. 2021 May;54:101888. doi: 10.1016/j.psychsport.2021.101888. Epub 2021 Jan 12. PMID 33633498
- [Background] Gjellesvik TI, Becker F, Tjonna AE, Indredavik B, Nilsen H, Brurok B, Torhaug T, Busuladzic M, Lydersen S, Askim T. Effects of High-Intensity Interval Training After Stroke (the HIIT-Stroke Study): A Multicenter Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Jun;101(6):939-947. doi: 10.1016/j.apmr.2020.02.006. Epub 2020 Mar 4. PMID 32145280
- [Background] Izquierdo MC, Lopes S, Teixeira M, Polonia J, Alves AJ, Mesquita-Bastos J, Ribeiro F. The Chester step test is a valid tool to assess cardiorespiratory fitness in adults with hypertension: reducing the gap between clinical practice and fitness assessments. Hypertens Res. 2019 Dec;42(12):2021-2024. doi: 10.1038/s41440-019-0316-5. Epub 2019 Aug 26. No abstract available. PMID 31451720
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Background] Montori VM, Guyatt GH. Intention-to-treat principle. CMAJ. 2001 Nov 13;165(10):1339-41. No abstract available. PMID 11760981
- [Background] Murawska-Cialowicz E, Wolanski P, Zuwala-Jagiello J, Feito Y, Petr M, Kokstejn J, Stastny P, Golinski D. Effect of HIIT with Tabata Protocol on Serum Irisin, Physical Performance, and Body Composition in Men. Int J Environ Res Public Health. 2020 May 20;17(10):3589. doi: 10.3390/ijerph17103589. PMID 32443802
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632
- [Background] Severo M, Santos AC, Lopes C, Barros H. [Reliability and validity in measuring physical and mental health construct of the Portuguese version of MOS SF-36]. Acta Med Port. 2006 Jul-Aug;19(4):281-7. Epub 2007 Jan 23. Portuguese. PMID 17328844
- [Background] Stergiou GS, Alpert BS, Mieke S, Wang J, O'Brien E. Validation protocols for blood pressure measuring devices in the 21st century. J Clin Hypertens (Greenwich). 2018 Jul;20(7):1096-1099. doi: 10.1111/jch.13294. PMID 30003697
- [Background] Sykes, K., & Roberts, A. (2004). The Chester step test-a simple yet effective tool for the prediction of aerobic capacity. Physiotherapy, 90(4), 183-188. https://doi.org/10.1016/j.physio.2004.03.008
- [Background] Tabata I. Tabata training: one of the most energetically effective high-intensity intermittent training methods. J Physiol Sci. 2019 Jul;69(4):559-572. doi: 10.1007/s12576-019-00676-7. Epub 2019 Apr 19. PMID 31004287
- [Background] Teques P, Calmeiro L, Silva C, Borrego C. Validation and adaptation of the Physical Activity Enjoyment Scale (PACES) in fitness group exercisers. J Sport Health Sci. 2020 Jul;9(4):352-357. doi: 10.1016/j.jshs.2017.09.010. Epub 2017 Sep 29. PMID 32768128
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Wijndaele K, Westgate K, Stephens SK, Blair SN, Bull FC, Chastin SF, Dunstan DW, Ekelund U, Esliger DW, Freedson PS, Granat MH, Matthews CE, Owen N, Rowlands AV, Sherar LB, Tremblay MS, Troiano RP, Brage S, Healy GN. Utilization and Harmonization of Adult Accelerometry Data: Review and Expert Consensus. Med Sci Sports Exerc. 2015 Oct;47(10):2129-39. doi: 10.1249/MSS.0000000000000661. PMID 25785929

DOCUMENTS (1):
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT04796532/ICF_000.pdf